CLINICAL TRIAL: NCT05856630
Title: A Randomized, Open-label, Parallel, Active-controlled Phase 1 Study to Compare Pharmacokinetics Pharmacodynamics and Safety of Goserelin Acetate Sustained-Release Microspheres for Injection (LY01022) With Zoladex® 10.8mg Following Single Administration in Patients With Prostate Cancer
Brief Title: Pharmacokinetics Pharmacodynamics and Safety of LY01022 in Patients With Prostate Cancer Compared With Zoladex® 10.8mg
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LY01022/CT-CHN-101
Record Dates: First submitted 2023-04-22; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Injections; Goserelin; Drug Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LY01022 (Experimental)
  Interventions: Drug: Goserelin Acetate Sustained-Release Microspheres for Injection
- Zoladex® (Active Comparator)
  Interventions: Drug: Zoladex 10.8 MG Drug Implant

INTERVENTIONS:
Drug: Goserelin Acetate Sustained-Release Microspheres for Injection — 10.8mg, Single dose, subcutaneously（SC）
  Other Names: LY01022
  Arms: LY01022
Drug: Zoladex 10.8 MG Drug Implant — 10.8mg, Single dose, subcutaneously（SC）
  Arms: Zoladex®

SUMMARY:
This is a randomized, open-label, Parallel, active-controlled phase I study. A total of 20-24 patients with locally advanced or metastatic prostate cancer will be randomized in a 1:1 ratio to receive a single injection of LY01022 10.8mg or Zoladex® 10.8mg. Blood samples will be collected to evaluate PK and PD profiles, and safety evaluation will be conducted as required in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Patients with locally advanced or metastatic prostate cancer suitable for endocrine therapy, including those who are suitable for endocrine therapy following radical therapy.
* Serum testosterone level ≥ 150 ng/dL (1.50 ng/mL or 5.2 nmol/L) at the screening visit.
* Life expectancy of at least 9 months.
* ECOG score of ≤ 2.
* Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L, platelet count ≥ 90 x 10^9/L, white blood cell count ≥ 3 x 10^9/L, hemoglobin ≥ 90 g/L.
* Total bilirubin (TBIL) ≤ 1.5×ULN, ALT and AST ≤ 3×ULN (or ≤ 5.0×ULN for patients with liver metastases).
* Creatinine clearance ≥50 mL/min at the screening visit.
* Subjects of childbearing potential must agree to use a reliable method of contraception with their female sexual partners during the study period and at least 6 months after the last administration.
* Patients who voluntarily sign an IRB-approved informed consent form before any trial-related activities, are willing to abide by the restrictions of the study, and complete the prescribed examinations.

Exclusion Criteria:

* Patients with prostate cancer who receive previous or ongoing endocrine therapy (surgical castration or other endocrine therapy including GnRH receptor agonists, GnRH receptor antagonists, anti-androgens, estrogens, megestrol acetate, etc.), except for patients with prostate cancer undergoing prostatectomy, radiotherapy or cryotherapy who have received neoadjuvant/adjuvant endocrine therapy for no more than 6 months and discontinued the above therapy more than 6 months before screening.
* Patients with confirmed or suspected hormone-resistant prostate cancer.
* Patients who have received prostatic surgery within 4 weeks prior to the first dose, or plan to receive major surgical treatment during the trial.
* Patients who have previously received hypophysectomy or adrenalectomy, or who have pituitary lesions or adrenal dysfunction.
* History of severe asthma, anaphylaxis, or severe urticaria and/or angioedema.
* Other cancer diseases diagnosed within 5 years before the screening visit, except for surgically removed basal or squamous cell carcinoma of the skin.
* History of the following medical histories within 6 months prior to the screening visit: stroke, transient ischemic attack (TIA), myocardial infarction, unstable angina, coronary revascularization, New York Heart Association (NYHA) class ≥ II cardiac insufficiency, severe unstable arrhythmia.
* Hypertensive patients with poor blood pressure control (SBP ≥ 160 mmHg or DBP ≥ 100 mmHg at the screening visit).
* Patients with type 1 diabetes or type 2 diabetes with poor glycemic control (glycosylated hemoglobin > 8% at the screening visit).
* Patients who have received treatment with 5-α reductase inhibitors (finasteride, dutasteride, enalidomide, epristeride, etc.) within 4 weeks before the first dose.
* Patients who are receiving coumarin anticoagulants at the screening visit.
* Have congenital long QT syndrome or QT/QTc interval prolongation (QTc ≥ 450 ms) at the screening visit; Or has received drugs that may prolong QT/QTc interval at the screening visit.
* Known to be allergic to the active ingredients or any excipients of GnRH agonists or bicalutamide.
* Patients who are seropositive for hepatitis B surface antigen (HBsAg), and must meet the following 2 conditions at the same time: 1. HBV DNA level: HBeAg-positive patients, HBV DNA ≥ 20,000 IU/ml [equivalent to 10^5 copies/mL]; HBeAg-negative patients, HBV DNA ≥ 2,000 IU/ml [equivalent to 10^4 copies/mL]; 2. ALT ≥ 2 x ULN);
* Patients who are seropositive for HIV antibody or HCV antibody.
* Alcoholics or drug abusers. Alcoholics are defined as drinking more than 14 units of alcohol per week within 3 months prior to the screening visit (1 unit = 350 mL beer, or 45 mL liquor, or 150 mL wine).
* Have participated in any clinical trials of investigational drugs or medical devices, and discontinued within 1 month before the screening visit.
* Other conditions considered unsuitable for enrollment by the investigator (such as spinal cord compression due to prostate cancer metastatic lesions of pyramid, pulmonary interstitial disease or other serious diseases).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Changes in plasma goserelin concentration after administration of LY01022 or Zoladex® | from baseline to Day 99

SECONDARY OUTCOMES:
Changes in serum testosterone concentration after administration of LY01022 or Zoladex® | from baseline to Day 99
Changes in serum luteinizing hormone (LH) concentration after administration of LY01022 or Zoladex® | from baseline to Day 99
Changes in serum follicle stimulating hormone (FSH) concentration after administration of LY01022 or Zoladex® | from baseline to Day 99
Adverse events throughout the study | from baseline to Day 99

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, China